CLINICAL TRIAL: NCT06502626
Title: Effects of Sprint Interval Training on Speed, Change of Direction and Running Performance Among Field Hockey Players.
Brief Title: Effects of Sprint Interval Training on Field Hockey Players.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0477
Record Dates: First submitted 2024-06-11; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Sports Physical Therapy
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sprint Interval Training (Experimental): Sprint interval training will be given for 4 weeks. Each week consisted of three training sessions, separated by at least one resting day. Participants will complete a 15-minutes warm up before training session. The Sprint interval training group consisted of 30 s sprints at near maximal effort, with three minutes of rest between each sprint. The training intensity of Sprint interval training sessions was evaluated subjectively during sessions. During the first week, the Sprint interval training group performed five sprints per session. The number of sprints then increased gradually, until a total of 10 sprints per session. When the number of sprints reached seven, subjects were given six minutes of rest midway through the training session
  Interventions: Other: Sprint Interval Training
- Regular Training (Other): Regular training will be done.
  Interventions: Other: Regular training

INTERVENTIONS:
Other: Regular training — performed their routine programs
  Arms: Regular Training
Other: Sprint Interval Training — Sprint interval training will be given for 4 weeks. Each week consisted of three training sessions, separated by at least one resting day. Participants will complete a 15-minutes warm up before training session. The Sprint interval training group consisted of 30 s sprints at near maximal effort, with three minutes of rest between each sprint. The training intensity of Sprint interval training sessions was evaluated subjectively during sessions. During the first week, the Sprint interval training group performed five sprints per session. The number of sprints then increased gradually, until a total of 10 sprints per session. When the number of sprints reached seven, subjects were given six minutes of rest midway through the training session
  Arms: Sprint Interval Training

SUMMARY:
Field hockey is a team sport that is played using sticks and balls. Player's motions are impromptu and determine how competitive matches are played. Athletes can enhance their performance through a variety of training regimens. "Sprint Interval Training," for short bursts of maximal or supramaximal exercise, is one type of training used to improve sports performance. During recovering intervals, participants alternate between passive rest or light to moderately hard work. In both skilled and novice players, Sprint interval training significantly increases anaerobic and aerobic performance. This study aims to determine the impact of sprint interval training on hockey player's running performance, speed, and direction changes.

DETAILED DESCRIPTION:
Field hockey is a team sport played with sticks and balls in which players' movements are spontaneous and dictate the fluctuating nature of competitive match play. A number of training programs are used to improve the performance of the athlete. One of the trainings that is used to enhance the performance of a sports person is "Sprint Interval Training" and it consists of short bursts of maximal or supramaximal exercise interspersed with passive rest or light to moderately intense exertion during rebound periods. Sprint interval training dramatically improves anaerobic and aerobic performance in both trained and untrained athletes. The aim of this study is to find the effect of sprint internal training on speed, change of direction and running performance among field hockey players.

A randomized controlled trial will be conducted at Pakistan Sports Academy, Lahore through non-probability convenience sampling technique on 28 players which will be allocated into both interventional and control group. Pre-training values of the players will be recorded by 20 m sprint test for speed, 505 Change of direction test for change of direction and 3000m time trial for running performance. Both groups will perform regular training. Sprint interval training will be given to Group A and regular training will be performed by Group B. Players will perform the training 3 times a week for 4 weeks and treatment evaluation will be done after 4 weeks. Data will be analyzed using SPSS software version 26. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years.
* Both males and females.
* Moderate level of training (Approximately 3 hours per week of activity).
* Playing experience of minimum 2 years.
* Being physically active in a self-reported manner (Approximately 150 minutes of physical activity weekly).

Exclusion Criteria:

* Systemic Conditions (unstable angina, systemic arterial hypertension, chronic obstructive pulmonary disease, diabetes mellitus, neoplasm, renal failure and sequelae of stroke).
* Any musculoskeletal issues that made it difficult to follow protocols or conduct testing.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
Speed | 10 months
  It will be assessed by 20m sprint test, values will be taken before and after the application of sprint interval training for the participants of both groups.
Change of direction | 10 months
  It will be assessed by 505 Change of direction test, values will be taken before and after the application of sprint interval training for the participants of both groups.
Running performance | 10 months
  It will be assessed by 3000m time trial, values will be taken before and after the application of sprint interval training for the participants of both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, T-DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports Academy, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No